CLINICAL TRIAL: NCT00134212
Title: Prospective, Randomized Study on Two Parallel Groups Comparing Dopexamine and Norepinephrine in Combination to Epinephrine Alone on Systemic and Pulmonary Hemodynamics, Gastric Mucosal Perfusion, and Oxidative Stress in Septic Shock
Brief Title: Dopexamine and Norepinephrine Compared With Epinephrine Alone in Septic Shock
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AFSSAPS 020193; LOC-H/01-08; CIC0203/008
Record Dates: First submitted 2005-08-22; First posted 2005-08-24 (Estimated); Last update posted 2006-01-02 (Estimated); Status verified 2005-12

CONDITIONS: Septic Shock
Keywords: Splanchnic perfusion, hepatic damage, oxidative stress.
MeSH Terms: conditions — Shock, Septic | interventions — dopexamine; Norepinephrine; Epinephrine

INTERVENTIONS:
Drug: Dopexamine and norepinephrine
Drug: Epinephrine

SUMMARY:
In septic shock, when volume resuscitation fails to restore mean arterial pressure, catecholamines such as dopamine, dobutamine, epinephrine, or norepinephrine are used, either alone or in combination. Although they allow hemodynamic success to be obtained, they can leave some regional blood flows impaired, especially the hepatosplanchnic perfusion, which contributes to multiple organ failure.

Dopexamine is a structural and synthetic analog of dopamine that exerts systemic and gut vasodilation and stimulates cardiac contraction. In experimental models, dopexamine has been shown to exert anti-inflammatory properties and to protect the hepatic ultra structure. The combination of dopexamine and norepinephrine could therefore constitute an interesting alternative in treating septic shock patients. This study will test the efficacy (on gastric mucosal blood flow, hepatic damage and oxidative stress) and safety of the combination of dopexamine and norepinephrine (compared to those of epinephrine alone) in the treatment of patients with septic shock.

DETAILED DESCRIPTION:
Objective: To compare the combination of dopexamine and norepinephrine with epinephrine alone on gastric mucosal blood flow (GMBF), hepatic damage and oxidative stress in septic shock.

Setting: Surgical intensive care unit in a university hospital.

Design: Prospective, randomized, controlled study on 2 parallel groups.

Patients: Adults fulfilling usual criteria for septic shock.

Interventions: Systemic hemodynamics, GMBF (laser-Doppler), plasma α-glutathione S-transferase, aspartate aminotransferase, alanine aminotransferase and malondialdehyde were assessed just before catecholamine infusion (T0), as soon as mean arterial pressure (MAP) reached 70-80 mmHg (T1), and 2 (T2) and 6 (T3) hours after T1. Drugs were titrated from 0.2 µg/kg/min with 0.2 µg/kg/min increments every 3 min for epinephrine and norepinephrine, and from 0.5 µg/kg/min with 0.5 µg/kg/min increments every 3 min for dopexamine.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years
* Informed consent
* Septic shock with:

  * evidence of infection;
  * at least 3 of the following criteria: temperature > 38°C or < 36.5°C; respiratory rate > 20 breaths per minute or PaCO2 < 32 mmHg or mechanical ventilation; heart rate > 90 beats/min; white blood cell count > 12,000/mm3 or < 4,000/mm3;
  * at least 2 of the following criteria: plasma lactate > 2 mmol/L or unexplained metabolic acidosis (pH < 7.3); hypoxemia defined by PaO2 < 70 mmHg at room air or a PaO2/FiO2 ratio < 280 mmHg (or < 200 mmHg if pneumonia was the source of sepsis) or need for mechanical ventilation; urine output < 30 mL/h for at least 2 hours despite a fluid challenge of at least 500mL; a platelet count < 100,000/mm3, a decrease of 50% from previous value, or unexplained coagulopathy (prothrombin time < 60% and elevated fibrin degradation products > 10 μg/mL);
  * systolic blood pressure < 90 mmHg despite an optimal volume loading defined by a pulmonary capillary wedge pressure > 12 mmHg.

Exclusion Criteria:

* Pregnant women
* Patients with a history of esophageal or gastric disease
* Patients with a history of esophageal or gastric surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2002-03; Study Completion 2004-06

PRIMARY OUTCOMES:
Gastric mucosal blood flow assessed using a laser-Doppler flowmeter

SECONDARY OUTCOMES:
Systemic and pulmonary hemodynamics: systolic, diastolic and mean arterial, right atrial, systolic, diastolic and mean pulmonary arterial, and pulmonary capillary wedge pressures
heart rate, stroke volume, cardiac output
systemic and pulmonary vascular resistances
arterial and venous blood gases and arterial lactate
alanine and aspartate amino transferases
bilirubin
α-glutathione S-transferase
nitric oxide and reactive oxygen species productions

CONTACTS AND LOCATIONS:
Overall Officials: Yannick Mallédant, MD, Study Director — Rennes University Hospital; Eric Bellissant, MD, PhD, Study Chair — Rennes University Hospital; Philippe Seguin, MD, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes University Hospital, Rennes, France

REFERENCES:
- [Background] Schmidt W, Hacker A, Gebhard MM, Martin E, Schmidt H. Dopexamine attenuates endotoxin-induced microcirculatory changes in rat mesentery: role of beta2 adrenoceptors. Crit Care Med. 1998 Oct;26(10):1639-45. doi: 10.1097/00003246-199810000-00012. PMID 9781719
- [Background] Tighe D, Moss R, Heywood G, al-Saady N, Webb A, Bennett D. Goal-directed therapy with dopexamine, dobutamine, and volume expansion: effects of systemic oxygen transport on hepatic ultrastructure in porcine sepsis. Crit Care Med. 1995 Dec;23(12):1997-2007. doi: 10.1097/00003246-199512000-00008. PMID 7497722
- [Derived] Seguin P, Laviolle B, Guinet P, Morel I, Malledant Y, Bellissant E. Dopexamine and norepinephrine versus epinephrine on gastric perfusion in patients with septic shock: a randomized study [NCT00134212]. Crit Care. 2006 Feb;10(1):R32. doi: 10.1186/cc4827. PMID 16507156